CLINICAL TRIAL: NCT01054677
Title: Swedish Antibiotic Nursing Home Trial
Acronym: SANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The national corporation of Swedish pharmacies, Apoteket AB (Unknown)
Responsible Party: Cecilia Stålsby Lundborg, Karolinska Institutet
Purpose: Health Services Research
Other Study IDs: dnr 03-070
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2003-05

CONDITIONS: Infections; Urinary Tract Infections
Keywords: Infections in nursing homes; especially urinary tract infections
MeSH Terms: conditions — Infections; Urinary Tract Infections

ARMS (2):
- Educational intervention on antibiotic prescribing (Experimental): The participants in this group received an educational intervention.
  Interventions: Behavioral: Educational intervention on antibiotic prescribing
- No educational intervention (No Intervention): The participants in this group did not receive the educational intervention

INTERVENTIONS:
Behavioral: Educational intervention on antibiotic prescribing — Small educational group sessions with nurses and physicians, feedback on prescribing, presentation of guidelines and written materials
  Arms: Educational intervention on antibiotic prescribing

SUMMARY:
Main aim and objective

The aim was to present the treatment of infectious diseases in elderly, especially in nursing homes and further to evaluate the effect of an intervention package aiming at improving treatment with antibiotics in Swedish nursing homes

Specific objectives

* Present the treatment patterns regarding infectious diseases, including gender aspects in elderly, especially in nursing homes.
* Through focus group discussions elucidate the decision making process in nursing homes and target the intervention.
* Based on the above information develop an educational intervention to contribute to the improvement of the prescribing of antibiotics in nursing homes
* Evaluate the effect of the intervention on quality of prescribing, knowledge and attitudes in relation to available guidelines

ELIGIBILITY:
Inclusion Criteria:

* nursing homes where residents have a common dining room and staff, and a self-assessed stable staff situation

Exclusion Criteria:

* specialised nursing homes or wards (e.g. oncology wards)

Age Groups: Child, Adult, Older Adult